CLINICAL TRIAL: NCT01166542
Title: Randomized, Double-blind, Multicenter Two-Stage Adaptive Phase 3 Study of Intravenous Administration of REOLYSIN (Reovirus Type 3 Dearing) in Combination With Paclitaxel and Carboplatin Versus the Chemotherapy Alone in Patients With Metastatic or Recurrent Squamous Cell Carcinoma of the Head and Neck Who Have Progressed on or After Prior Platinum-Based Chemotherapy
Brief Title: Efficacy Study of REOLYSIN® in Combination With Paclitaxel and Carboplatin in Platinum-Refractory Head and Neck Cancers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oncolytics Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REO 018
Record Dates: First submitted 2010-07-13; First posted 2010-07-21 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Carcinoma, Squamous Cell of the Head and Neck
Keywords: carcinoma; squamous cell; head; neck; REOLYSIN (Reovirus Type 3 Dearing); chemotherapy; Carboplatin; Paclitaxel; metastatic; recurrent
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma; Neoplasm Metastasis; Recurrence | interventions — reolysin; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- REOLYSIN, paclitaxel, carboplatin (Active Comparator)
  Interventions: Biological: REOLYSIN; Drug: Carboplatin; Drug: Paclitaxel
- placebo, paclitaxel, carboplatin (Placebo Comparator)
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Biological: REOLYSIN — 3E10 TCID50, 1 hour intravenous infusion, administered on Days 1, 2, 3, 4 and 5 of a 21 day cycle
  Other Names: reovirus serotype 3 Dearing Strain
  Arms: REOLYSIN, paclitaxel, carboplatin
Drug: Carboplatin — 5 AUC mg/mL min, 30 min intravenous infusion, given on Day 1 of a 21 day cycle
Drug: Paclitaxel — 175 mg/m2, 3 hour intravenous infusion, given on Day 1 of a 21 day cycle
Drug: Placebo — Placebo
  Arms: placebo, paclitaxel, carboplatin

SUMMARY:
The purpose of this Phase 3 study is to evaluate overall survival and progression free survival following intravenous administration of REOLYSIN (Reovirus Serotype 3 Dearing) in combination with paclitaxel and carboplatin versus chemotherapy treatment alone, in patients with metastatic or recurrent Squamous Cell Carcinoma of the Head and Neck.

DETAILED DESCRIPTION:
Squamous cell carcinoma of the head and neck is the sixth most common cancer in the world. More than 50% of patients diagnosed with advanced regional disease will relapse locally or at distant sites. Initial therapeutic options include irradiation, surgery and chemotherapy. The most commonly used agents are cisplatin and carboplatin, generally in combination with 5-FU or a taxane. Erbitux has been approved for use in first-line with radiation and in second-line as monotherapy. Only about a third of the patients will respond to first-line platinum-based therapy and the median overall survival is about 6-9 months.

Preliminary assessment of a Phase 1-2 study conducted in the UK investigating the combination of REOLYSIN, carboplatin and paclitaxel suggested that patients with head and neck carcinomas may represent a group of patients in whom this treatment combination is active. Studies have also shown that paclitaxel and carboplatin combination therapy may be effective in head and neck cancers, even in heavily pretreated patients and those resistant to previous treatment. These results strongly support the utility of the carboplatin/paclitaxel combination as a control arm for salvage therapy in platinum refractory patients, a patient group with few and poor treatment options and with no gold standard therapy.

This Phase 3 study is designed to compare response rates following intravenous administration of REOLYSIN (Reovirus Type 3 Dearing) in combination with paclitaxel and carboplatin versus chemotherapy treatment alone, in patients with metastatic or recurrent Squamous Cell Carcinoma of the Head and Neck.

Overall survival is a primary endpoint of this trial. Patients will be clinically evaluated after each course of treatment and radiologically every 6 weeks on and after treatment. The safety of the paclitaxel and carboplatin with intravenous blinded placebo or intravenous blinded REOLYSIN will also be assessed.

ELIGIBILITY:
Inclusion Criteria: Each patient MUST:

* have recurrent or metastatic (R/M) histologically confirmed squamous cell carcinoma (SCC) of the head and neck (oropharynx, oral cavity, larynx, hypopharynx) or squamous cell nasopharynx cancer (NPC) with distal metastasis(es) and no secondary cancers (Patients with NPC without distal metastasis(es) or with undifferentiated NPC are not eligible).
* have at least one lesion that is measurable by computed tomography or magnetic resonance imaging (Lesions persisting in previously treated radiation fields are considered not evaluable for response except if representing a relapse in a mucosal or nodal lesion that previously demonstrated a complete response. Any new lesion within the previous radiation fields is acceptable for determination of response and/or progression).
* have completed first line chemotherapy for R/M SCCHN which progressed on or within 190 days following the completion of platinum or platinum-based chemotherapy.
* have no continuing acute toxic effects (except alopecia) of any prior radiotherapy, chemotherapy, or surgical procedures. Any surgery involving the SCC for which the patient is being treated (except biopsies) must have occurred at least 28 days prior to study enrollment.
* have received no chemotherapy, radiotherapy, immunotherapy or hormonal therapy within 28 days.
* have ECOG Performance Score of ≤ 2.
* have life expectancy of at least 3 months.
* absolute neutrophil count (ANC)≥ 1.5 x 10^9/L ; platelets ≥100 x 10^9/L]; hemoglobin ≥9.0 g/dL; serum creatinine ≤1.5 xULN; bilirubin ≤1.5 x ULN; AST/ALT ≤2.5 x ULN.
* negative pregnancy test for females with childbearing potential.
* Be wiling and able to comply with scheduled visits, the treatment plan, and laboratory tests.

Exclusion Criteria: No patient may:

* receive concurrent therapy with any other investigational anticancer agent while on study.
* have been treated with a taxane for SCCHN.
* have current -- or with a history of -- brain metastases because of their poor prognosis and because of the frequent development of progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* be on chronic immunosuppressive therapy or have known HIV infection or active hepatitis B or C.
* be a pregnant or breast-feeding woman. Female patients of childbearing potential must agree to use effective contraception, be surgically sterile, or be postmenopausal. Male patients must agree to use effective contraception or be surgically sterile. Barrier methods are a recommended form of contraception.
* have clinically significant cardiac disease (New York Heart Association, Class III or IV) including, but not limited to, pre-existing arrhythmia, uncontrolled angina pectoris, or myocardial infarction within 1 year prior to study entry.
* have dementia or any altered mental status that would prohibit informed consent.
* have any other acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Principal Investigator, would make the patient inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Overall survival | every 3 months until death.

SECONDARY OUTCOMES:
Progression-free survival | Assessed every 6 weeks until disease progression or death.
Objective response (complete response (CR) + partial response (PR)) rate and duration | Evaluation of response is conducted every 6 weeks on and after study. Duration of objective response is measured from the time measurement criteria are first met for CR or PR until recurrent or progressive disease is objectively documented.
Number of participants with adverse events as a measure of safety and tolerability of REOLYSIN when administered in combination with paclitaxel and carboplatin. | Within 30 days of the last dose of REOLYSIN.
Compare Best % Tumor Specific Response in loco-regional disease and/or metastatic disease for the treatment regimens in the study population | Assessed every 6 weeks until disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: James A Bonner, MD, Principal Investigator — University of Alabama at Birmingham, Birmingham, AB, US; Kevin Harrington, MBBS MRCP FRCR, Principal Investigator — The Royal Marsden Hospital, London, UK; Jan Vermorken, MD, PhD, Principal Investigator — University Hospital, Antwerp, Belgium
Locations (77):
- United States (21):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Oncology Associates, Tucson, Arizona
  - Providence Health and Services, Burbank, California
  - Wilshire Oncology Medical Group, Corona, California
  - BMS Physician Practice, A Medical Corporation DBA Medical Oncology Care Associates, Orange, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Pasco Hernando Oncology Associates, PA, New Port Richey, Florida
  - Emory University - Winship Cancer Institute, Altanta, Georgia
  - Alexian Brothers Hospital Network, Elk Grove Village, Illinois
  - Mary Bird Perkinds Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Montefiore Medical Center, The Bronx, New York
  - Case Comprehensive Cancer Center, University Hospitals Case Medical Center, Cleveland, Ohio
  - Mercy Cancer Center, Toledo, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Oncology- Sammons Cancer Center, Dallas, Texas
  - Cancer Therapy and Research Center at UTHSCSA, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Columbia Basin Hematology and Oncology, Kennewick, Washington
- Belgium (3):
  - ZNA Middelheim, Antwerp
  - University Hospital Antwerp, Edegem
  - Universitair Ziekenhuis Brussel, Jette
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Juravinski Cancer Center, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Hopital Notre-Dame, Montreal, Quebec
- France (3):
  - Hopital Saint-André / Service d'Oncologie-Radiothérapie, Bordeaux
  - Centre Antoine Lacassagne / Oncologie Médicale, Nice
  - Institut Curie / Département d'Oncologie Médicale, Paris
- UKE Hamburg, Hamburg, Germany
- Attikon University Hospital, Athens, Greece
- Hungary (5):
  - Fovarosi Onkormanyzat Uzsoki Utcai Kórház, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Pecsi Tudomanyegyetem, Pécs
  - Szegedi Tudományegyetem, Szegedi
  - Markusovszky Korhaz, Szombathely
- Italy (4):
  - Ufficio Sperimentazioni Cliniche c/o S.C. Oncologia Medica, Cuneo
  - Fondazione IRCCS Istituto Nazionale del Tumori, Milan
  - Ospedale San Paolo - Oncologia Medica, Milan
  - University Hospital in Modena, Modena
- Poland (4):
  - Centrum Onkologii - Instytyt im.M.Skłodowskiej-Curie, Krakow
  - Wojewódzki Szpital Specjalistyczny im. M.Kopernika, Lodz
  - Szpital MSWiA - Centrum Onkologi, Olsztyn
  - Wielkopolskie Centrum Onkologii, Poznan
- Russia (14):
  - State Health Care Institution "Arkhangelsk Regional Clinical Oncology Dispensary", Arkhangelsk
  - Regional State Health Care Institution "Belgorod Oncology Dispensary", Belgorod
  - State Health Care Institution "Chelyabinsk Regional Oncology Dispensary", Chelyabinsk
  - State Health Care Institution "Republican Clinical Oncology Dispensary of Ministry of Health of the Republic of Tatarstan", Kazan'
  - State Budgetary Health Care Institution "Clinical Oncology Dispensary #1" of Krasnodar Region Health Care Department, Krasnodar
  - Regional Budgetary Health Care Institution "Kursk Regional Oncology Dispensary" of Health Care Committee of Kursk region, Kursk
  - Federal State Budgetary Institution "Medical Research Radiology Center" of Ministry of Public Health and Social Development of Russian Federation, Obninsk, Obninsk
  - Federal State Budgetary Institution "N. N. Petrov Oncology Research Institute" of Ministry of Public Health and Social Development of the Russian Federation, Saint Petersburg
  - Federal State Budgetary Institution "Russian Research Centre of Radiology and Surgery technologies" of Ministry of Public Health and Social Development of the Russian Federation, Saint Petersburg
  - St.Petersburg State Health Care Institution City Clinical Oncology Dispensary", Saint Petersburg
  - State Health Care Institution "Oncology Dispensary №2" of Krasnodar Region Health Care Department, Sochi
  - State Health Care Institution "Tula Regional Oncology Dispensary", Tula
  - State Budgetary Healthcare Institution "Republic Clinical Oncology Dispensary Ministry of Health of Bashkortostan", Ufa
  - State Budgetary Health Care Institution of the Yaroslavl region "Regional Clinical Oncological Hospital", Yaroslavl
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- Spain (7):
  - Hospital Vall D'Hebron, Barcelona
  - Instituto Catlan de Oncologia (ICO) - Hospital Duran i Reynals, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Instituto Catlan de Oncologia (ICO) - Hospital Germans Trias I Pujol, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital de Navarra, Pamplona
- United Kingdom (9):
  - Beatson West of Scotland Cancer Center, Glasgow
  - Royal Surrey County Hospital, Guildford
  - St. James's University Hospital, Leeds
  - Guy's and St. Thomas Hospital, London
  - The Royal Marsden Cancer Center, Fulham Road branch, London
  - Clatterbridge Centre for Oncology NHS Foundation Trust, Metropolitan Borough of Wirral
  - The Royal Marsden Cancer Center, Sutton Branch, Sutton
  - Musgrove Park Hospital, Taunton
  - The Velindre Hospital, Whitchurch